CLINICAL TRIAL: NCT04005443
Title: Molecular Imaging Exploration of Ocular Angiogenic Activityand Evaluation of Its Interest in the Therapeutic Follow-upof Patients With AMD (Age-related Macular Degeneration)
Brief Title: Molecular Imaging Exploration of Ocular Angiogenic Activity and Evaluation of Its Interest in the Therapeutic Follow-up of Patients With AMD (Age-related Macular Degeneration)
Acronym: DMLA-RGD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-06; 2019-000946-37 (EudraCT Number)
Record Dates: First submitted 2019-06-20; First posted 2019-07-02 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Radiopharmaceuticals

STUDY DESIGN:
Intervention Model Description: In this study, two 68Ga-NODAGA-RGD PET scans will be performed for each patient included :
  * The first PET will be carried out within a maximum of one month following the assessment initial ophthalmologic including OCT and measurement of visual acuity (M0);
  * The second PET scan will be performed at the same time as the ophthalmic assessment including OCT and measurement of visual acuity (at M4), before the 5th intraocular injection antiangiogenic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET at 68Ga-NODAGA-RGD (Other): The first PET scan will be performed within a maximum of one month following the initial ophthalmologic assessment including OCT and measurement of visual acuity (M0);
  Interventions: Other: radiopharmaceutical

INTERVENTIONS:
Other: radiopharmaceutical — his study will consist of a monthly intra-ocular injection of antiangiogenic and a follow-up ophthalmological consultation with OCT and visual acuity score

SUMMARY:
The main objective of this pilot study is to evaluate the ability of 68Ga-NODAGA-RGD PET imaging to demonstrate, in patients with unilateral AMD, a molecular therapeutic response to intraocular antiangiogenic injections at the end of the first phase. induction (after 3 months of treatment).

DETAILED DESCRIPTION:
To date, no functional imaging modality has been validated to assess the level angiogenic activity of choroidal neovascularization in AMD, while the therapeutic use of antiangiogenic agents is almost systematically in the form of intraocular injections.

The therapeutic response is observed anatomically and functionally only after 6 months of treatment. Several arguments in the literature suggest that the therapeutic response occurs earlier at the molecular level, as soon as the induction phase is complete (after 3 months of treatment). The main objective of this pilot study is to evaluate the ability of 68Ga-NODAGA-RGD PET imaging to demonstrate, in patients with unilateral AMD, a molecular therapeutic response to intraocular antiangiogenic injections at the end of the first phase. induction (after 3 months of treatment).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, membership of a social security scheme. Signature of informed consent,
* Subject presenting AMD with unilateral involvement, involving at least 1 Choroidal neovascularization objectified in OCT, naive to any treatment antiangiogenic.
* Initial assessment including at least OCT and measurement of visual acuity, dating from maximum 1 month at the time of PET 68Ga-NODAGA-RGD.

Exclusion Criteria:

* Pregnant or breastfeeding women, as a result of radiation protection.
* Subjects under 18 years of age and / or not affiliated to a social security scheme.
* Subjects with AMD with bilateral involvement.
* Subjects with AMD without a focus of neovascularization objectified by the classic diagnostic battery.
* Subjects having already been treated with antiangiogenic therapy.
* Subjects with any other ophthalmological pathology. Monophthalmic subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-02 (Actual); Primary Completion 2024-06-02 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of the signal intensity ratios of the AMD eye / contralateral eye TEP (SUVmax) signal | 7 months
  Images from the 68Ga-NODAGA-RGD PET scan will be interpreted without results of other examinations and clinical history. Two experienced nuclear physicians unfamiliar with the results of the initial balance sheet examinations will complete a grid listing the quantification of the 68Ga-NODAGA-RGD (SUVmax) signal measured in each eye of each patient.
  The signal intensity ratios of the AMD eye / contralateral eye TEP (SUVmax) signal at M0 and M4 will be compared by a comparison test of paired averages.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Garrido Pradalie, Study Director — Assistance Publique-Hôpitaux de Marseille
Locations (1):
- APHM, Marseille, France